CLINICAL TRIAL: NCT01252524
Title: Effect of Calcium Polycarbophil on Type II Diabetes Mellitus Control: a Randomized Double-blind Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Tae Joon Lee, Clinical Associate Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-0422
Record Dates: First submitted 2010-11-05; First posted 2010-12-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes Mellitus Type II
Keywords: diabetes mellitus; fiber; glycemic control; calcium polycarbophil
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — calcium polycarbophil; Psyllium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): A placebo tablet PO TID before each meal with 8 oz of water for 6 months.
  Interventions: Drug: Placebo
- Calcium polycarbophil (Experimental): Calcium polycarbophil 625 mg PO TID before each meal with 8 oz of water for 6 months
  Interventions: Drug: Calcium polycarbophil

INTERVENTIONS:
Drug: Placebo — Placebo tablet po TID before each meal with 8 oz of water for 6 months
  Arms: Placebo
Drug: Calcium polycarbophil — calcium polycarbophil 625 mg po TID before each meal with 8 oz water for 6 months
  Other Names: Konsyl; Fibercon
  Arms: Calcium polycarbophil

SUMMARY:
The purpose of this study is to determine whether a form of fiber if effective in improving the treatment of type 2 diabetes. Measurements of other possible medical benefits will include blood pressure, cholesterol, weight, and the number/dosage of medications used for diabetes, hypertension, and high cholesterol.

DETAILED DESCRIPTION:
There have been several publications in the medical literature linking the use of various types of fiber and the beneficial effects on lipid panel, glycosylated hemoglobin A1c, weight, blood pressure, and cardiovascular events in patients with type 2 diabetes mellitus or those at risk for diabetes1-5. Most of these studies utilize fiber sources from dietary food intake or psyllium.

However, diet modification and psyllium intake are difficult for patients to comply on daily basis and many patients do not continue to follow through on these interventions.

Polycarbophil is a bulk forming agent which is used for similar indications as psyllium for the treatment of constipation and irritable bowel syndrome. Because polycarbophil comes in oral tablets and capsules, patients may adhere to regular intake better compared to psyllium. However, it is unknown whether polycarbophil has similar beneficial properties compared to psyllium and other fiber types. Taking polycarbophil prior to each meal may improve diabetes control by allowing patients to have smaller meals and decrease the absorption rate of carbohydrates in the intestine.

The goal of this study is to determine whether taking calcium polycarbophil (also known as over-the-counter FiberconTM) regularly will improve the diabetes control. The proposed study will be a randomized, controlled, and double-blinded trial involving adult patients with type 2 diabetes mellitus. A total of 50 patients will be randomized to receive either calcium polycarbophil or placebo from the Family Medicine Center at East Carolina University and followed over 6 months. The primary outcome of the trial will be glycosylated hemoglobin A1c. Secondary outcome measures will include weight, blood pressure, and cholesterol level. Additional secondary outcome measures are the number and dosages of medications for diabetes mellitus, hypertension, and hyperlipidemia.

The potential benefits of this study include improved control of diabetes mellitus, hypertension, and hyperlipidemia, reflected by the improved outcomes mentioned above. Because calcium polycarbophil (FiberconTM) is a commonly used over-the-counter fiber product for constipation, and the dosage used in this study is well within the typical use recommended by the manufacturers, the potential adverse effects of this product is thought to be identical to that described for FiberconTM. Patients will receive their usual medical care by their own primary physicians regardless of their participation in this study. After the randomization to the intervention or the control group, the study team will only monitor the outcome measures and will not alter the medical care that the patients receive.

Study title:

Effects of calcium polycarbophil on type II diabetes mellitus control: a randomized double-blinded study.

Patient population:

East Carolina University Family Medicine Center (ECU FMC) outpatient clinic patients Age above 18 Diagnosed with type II diabetes mellitus (DM) for at least 24 months. At least 4 office visits within the past 24 months for DM follow up at ECU FMC or Geriatrics Center.

Hgb A1c within the past six months of 8% to 10%.

Exclusion criteria:

Dementia diagnosis or other psychiatric diagnoses that preclude the patient from being able to consent for this study by him/herself.

Already taking fiber supplementation (polycarbophil, psyllium, methylcellulose) Severe problems with previous use of fiber supplementation (i.e. fecal impaction) Dysphagia or other swallowing disorders (unable to swallow pills or 8 oz of water) Pregnancy during the study period

Consent:

Will be obtained from the patients for the study and HIPAA.

Study design:

Randomize 50 patients to intervention or placebo:

Intervention: 25 patients to receive calcium polycarbophil 625mg po TID before each meal with 8 oz glass of water for 6 months.

Placebo control: 25 patients to receive placebo po TID before each meal with 8 oz glass of water for 6 months.

Total of 50 participants projected from the following power calculation:

Assuming a difference between groups in HbA1c of 0.5%, a standard deviation of 0.5, a power of 80% and an alpha of 0.05, an estimated 18 patients in each group (n = 36 pts) will be needed to detect a difference. Assuming a 25% dropout rate, the goal of 25 patients in each group (n=50 pts) will be needed.

Patients, primary physicians, and the researchers will be blinded to therapy versus placebo. Randomization will be performed by the ECU FM pharmacist who will open a sealed envelope which will indicate whether the patient will receive the interventional medication or placebo. The tablets will be dispensed by the pharmacist without informing the patient, physicians, or research team member as to which group the patient was randomized.

All patient will continue with their usual DM care. The patients must follow up at 3 months and 6 months.

A research team member will perform telephone follow up at 1 week, 1 month, and 3 months for adverse events and compliance.

The outcomes will be analyzed by intention to treat analysis and analysis using patients who are compliant with the trial protocol.

Primary outcome:

HgbA1c at the time of enrollment, 3 months, and 6 months.

Secondary outcome:

Data will be gathered at the time of enrollment, 3 months, and 6 months:

Weight Blood Pressure Number and dosage of medications for diabetes, hypertension, and hyperlipidemia Serum LDL, HDL, triglycerides, total cholesterol Patient compliance with the study medication Adverse events including GI discomfort, constipation, excessive flatulence, fecal impaction, diarrhea, nausea, vomiting, hypoglycemia, etc.

Potential adverse events:

Side effects of Polycarbophil (MicroMedex 2.0): Abdominal fullness, flatus, vomiting, stomach cramps. Systemic adverse effects are not expected since calcium polycarbophil is not absorbed

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Diagnosed with type II diabetes mellitus for at least 24 months
* At least 4 office visits within the past 24 months for diabetes mellitus follow up at ECU Family Medicine Center
* Hemoglobin A1c within the past six months between 8% to 10%

Exclusion Criteria:

* Dementia diagnosis or other psychiatric diagnoses that preclude the patient from being able to consent for this study by him/herself
* Already taking fiber supplementation (polycarbophil, psyllium, methylcellulose)
* Severe problems with previous use of fiber supplementation
* Dysphagia or other swallowing disorders, preventing the subject from swallowing pills or 8 oz of water
* Pregnancy during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c from baseline | Enrollment, 3 months, 6 months
  Change in hemoglobin A1c will be measured during these time intervals to determine the effects of polycarbophil on diabetes mellitus control.

SECONDARY OUTCOMES:
Weight | Baseline, 3 months, 6 months
Blood Pressure | Baseline, 3 months, 6 months
Number and dosage of medications for DM, HTN, and hyperlipidemia | Baseline, 3 months, 6 months
Serum LDL, HDL, triglycerides, total cholesterol | Baseline, 3 months, 6 months
Adverse outcomes | 3 months, 6 months
  GI discomfort, constipation, excessive flatulence, fecal impaction, diarrhea, nausea, vomiting, hypoglycemia, other reported side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Tae J Lee, MD, CMD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University Family Medicine Center, Greenville, North Carolina, United States

REFERENCES:
- [Background] Chandalia M, Garg A, Lutjohann D, von Bergmann K, Grundy SM, Brinkley LJ. Beneficial effects of high dietary fiber intake in patients with type 2 diabetes mellitus. N Engl J Med. 2000 May 11;342(19):1392-8. doi: 10.1056/NEJM200005113421903. PMID 10805824
- [Background] Vuksan V, Jenkins DJ, Spadafora P, Sievenpiper JL, Owen R, Vidgen E, Brighenti F, Josse R, Leiter LA, Bruce-Thompson C. Konjac-mannan (glucomannan) improves glycemia and other associated risk factors for coronary heart disease in type 2 diabetes. A randomized controlled metabolic trial. Diabetes Care. 1999 Jun;22(6):913-9. doi: 10.2337/diacare.22.6.913. PMID 10372241
- [Background] Rodriguez-Moran M, Guerrero-Romero F, Lazcano-Burciaga G. Lipid- and glucose-lowering efficacy of Plantago Psyllium in type II diabetes. J Diabetes Complications. 1998 Sep-Oct;12(5):273-8. doi: 10.1016/s1056-8727(98)00003-8. PMID 9747644
- [Background] Ziai SA, Larijani B, Akhoondzadeh S, Fakhrzadeh H, Dastpak A, Bandarian F, Rezai A, Badi HN, Emami T. Psyllium decreased serum glucose and glycosylated hemoglobin significantly in diabetic outpatients. J Ethnopharmacol. 2005 Nov 14;102(2):202-7. doi: 10.1016/j.jep.2005.06.042. Epub 2005 Sep 8. PMID 16154305
- [Background] Ylonen K, Saloranta C, Kronberg-Kippila C, Groop L, Aro A, Virtanen SM; Botnia Dietary Study. Associations of dietary fiber with glucose metabolism in nondiabetic relatives of subjects with type 2 diabetes: the Botnia Dietary Study. Diabetes Care. 2003 Jul;26(7):1979-85. doi: 10.2337/diacare.26.7.1979. PMID 12832299